CLINICAL TRIAL: NCT04050631
Title: In Hospital Maternal Cardiac Arrests: Highlighting the Importance of the First 5 Minutes.
Brief Title: Critical Delays in Cardiopulmonary Resuscitation During Simulated Obstetric Crisis: a Prospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KidSIM Simulation Program (Network)
Responsible Party: Sponsor
Other Study IDs: REB19-0042
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Maternal Death During Childbirth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- L&D team: the first responders on L&D floor including : anesthesia, nurses and OBGYN
  Interventions: Behavioral: maternal arrest simulation on L&D floor

INTERVENTIONS:
Behavioral: maternal arrest simulation on L&D floor — AFE on L&D

SUMMARY:
Maternal cardiac arrest is underreported and continues to occur at rate of 1:20,000 pregnancies. Despite being predominantly younger patients, survival rates among pregnant women are poor with one case series reporting a survival rate of 6.9%. Resuscitation of a pregnant women can be challenging when compared to non-pregnant adults. Aggressive maneuvers (perimortum cesarean section) and multidisciplinary team efforts are required because of the anatomical and physiological changes associated with pregnancy, in addition to taking care of two patents (mother and fetus). The first 5 minutes from the onset of cardiac arrest are the most crucial in terms of neonatal survival. In maternal deaths involving acute cardiac arrest, advanced cardiac life support (ACLS) must be rapidly administered. Previous work suggests deficits in cardiac arrest care during maternal cardiac arrest. The current literature fails to adequately quantify the severity, timing and frequency of errors made during maternal cardiac arrest care amongst interprofessional healthcare teams.

The primary goal of this study is to characterize the quality of actions by first responders during simulated in-hospital maternal medical emergencies. Specific objectives are:

1. to examine critical delays by measuring the median duration of the interval between when a resuscitation maneuver was indicated and when it was initiated by first responders ( nursing staff at L&D attending the patient).
2. to describe the type and frequency of resuscitation errors identified as deviations from AHA guidelines during obstetric cardiac arrest. By addressing this gap in the literature, we hope to highlight areas of future education and/or innovation aimed at improving performance during maternal cardiac arrest care.

DETAILED DESCRIPTION:
The investigators are planning to conduct a pilot descriptive study involving Foothill Medical Centre (FMC), Calgary. Research ethics approval will be obtained. The trial will also be registered at clinicaltrials.gov

The sessions will take place at the labor and delivery floor (L&D) simulation lab at FMC. The proposed time for study completion is 18 months. No follow up is required for this study. The data will be collected by one of the investigators (Dr. Fatemah Qasem). In addition, the participants performance will be video recorded for further data collection and revision by the investigator team.

On the day of the simulation session, the participants will be pre-briefed to the simulation room, mannequin, and the equipment but will be naïve to the simulation scenario. The simulation scenario will involve amniotic fluid embolism (AFE) in a term pregnant parturient with singleton pregnancy. The patient will have a working epidural catheter in situ for labor analgesia and an 18G IV line. The parturient will develop cardiopulmonary collapse due to AFE requiring ACLS.

The scenario will be scripted by investigator team members. The same scenario will be used at both centers (FMC and RGH). The script will include the initial clinical vignette; vital signs; patient weight; laboratory values; planned changes in clinical status, including what and when decompensations should occur (eg, 4 minutes into scenario, the patient will progress to pulseless VT); and planned responses to actions by participants. Time 0 will be referred to the onset of the decompensation. For maintaining realism, little interaction will occur between participants and evaluators. If no one remembers to call the code team, then the emergency is managed with only L&D staff. Although the primary focus of this study is to assess the quality of resuscitation delivered by first responders before the code team's arrival, the exercise will also allow to assess the resuscitation skills of obstetric care unit team. The scenario will end at skin incision for delivery of the fetus. Thirty minutes will be used for debriefing time as part of the hospital staff education. Data collected during the debriefing, and discussion points will used for quality improvement purposes and will not be used as part of the study results.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric healthcare providers: including: nurses, nurse practitioners, respiratory therapists and residents (obstetric and anesthesia)
* Basic Life Support (BLS) or Advanced Cardiac Life Support (ACLS) certification within the past two years;

Exclusion Criteria:

* Not BLS certified.
* Participant refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care providers at L&D floor : Anesthesia, OBGYN, Nurses
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes will be the median duration of the interval between when a resuscitation maneuver is indicated and when it will be initiated by first responders. | 10/ minutes
  oxygenation
The primary outcomes will be the median duration of the interval between when a resuscitation maneuver is indicated and when it will be initiated by first responders. | 100-120/minutes
  chest compressions
The primary outcomes will be the median duration of the interval between when a resuscitation maneuver is indicated and when it will be initiated by first responders. | minutes
  defibrillation
The primary outcomes will be the median duration of the interval between when a resuscitation maneuver is indicated and when it will be initiated by first responders. | 5 minutes
  time to incision

SECONDARY OUTCOMES:
Quality of CPR | 15 mins
  Depth
Quality of CPR | 15 minutes
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cheng, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada

REFERENCES:
- [Background] Campbell TA, Sanson TG. Cardiac arrest and pregnancy. J Emerg Trauma Shock. 2009 Jan;2(1):34-42. doi: 10.4103/0974-2700.43586. PMID 19561954
- [Background] Dijkman A, Huisman CM, Smit M, Schutte JM, Zwart JJ, van Roosmalen JJ, Oepkes D. Cardiac arrest in pregnancy: increasing use of perimortem caesarean section due to emergency skills training? BJOG. 2010 Feb;117(3):282-7. doi: 10.1111/j.1471-0528.2009.02461.x. PMID 20078586
- [Background] Yeomans ER, Gilstrap LC 3rd. Physiologic changes in pregnancy and their impact on critical care. Crit Care Med. 2005 Oct;33(10 Suppl):S256-8. doi: 10.1097/01.ccm.0000183540.69405.90. PMID 16215345